CLINICAL TRIAL: NCT05859087
Title: The Feasibility of Providing Family Planning Counseling Services for Women With Chronic Medical Conditions in an Inpatient Setting
Brief Title: Family Planning Counseling for Women With Chronic Medical Conditions in an Inpatient Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High attrition.
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, Ryan Spielvogel, Principal Investigator, Sutter Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Family14_SIMR_Spielvogel
Record Dates: First submitted 2023-04-24; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Chronic Disease
Keywords: Contraception; Access to Contraception; Health Inequities; Acute Care Setting; Inpatient
MeSH Terms: conditions — Chronic Disease | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: 1:1:1 randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bedside Family Planning Counseling (Experimental): Patient is screened for pregnancy intention and then has a bedside family planning counseling session with the investigator taking into account pregnancy intention, medical conditions, medications, and previous contraception used. At the end of the conversation, if patient is desiring contraception, the patient is offered three contraception options (as appropriate for their medical conditions and paid for as part of the study) to be initiated prior to discharge: Etonogestrel implant, medroxyprogesterone 150 mg IM injection, or a year's supply of oral contraception pills.
  Interventions: Behavioral: Counseling
- Flyer (Experimental): Patient is given a flyer that recommends they discuss pregnancy intention and contraception with their OB/GYN or primary care physician.
  Interventions: Behavioral: Flyer
- Routine care (No Intervention): Patients receive a deception consent so as not to influence them by the consent process. Consent states that the purpose of the project is to study patterns of birth control usage of women admitted to the hospital. Patient is not given any further intervention.

INTERVENTIONS:
Behavioral: Counseling — Bedside pregnancy intention screening and family planning counseling with offer of bedside contraception initiation.
  Arms: Bedside Family Planning Counseling
Behavioral: Flyer — Handing flyer to patient that discusses the importance of talking with their doctor about pregnancy intention and contraception use.
  Arms: Flyer

SUMMARY:
Women with chronic medical conditions have been found in multiple studies to use birth control less often compared to women without chronic medical conditions. The investigators hypothesized that approaching women with chronic medical conditions who were admitted to the hospital and having a bedside conversation about pregnancy intention and counseling regarding birth control usage along with offering to start birth control before discharge would increase the use of birth control in this population. As a separate intervention, the investigators hypothesized that having a brief conversation with the participants and then giving them a flyer that recommended talking with their doctor about birth control could also increase the use of birth control in this population.

ELIGIBILITY:
Inclusion Criteria:

* Currently admitted to the hospital
* Has one or more qualifying chronic medication conditions listed in their chart (hypertension, obesity with BMI>35, diabetes, current or history of breast cancer, rheumatoid arthritis, sickle cell disease, or lupus)

Exclusion Criteria:

* Currently pregnant
* Using surgical or non-surgical contraception
* Immediately post-partum or admitted to the gynecology service
* Non-English speaking
* Non-verbal or too ill to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Contraception use - 3 months | 3 months
  Number of patients using contraception 3 months post discharge as ascertained by telephone interview.
Pregnancy - 3 months | 3 months
  Number of pregnancies 3 months post discharge as ascertained by telephone interview.
Contraception use - 12 months | 12 months
  Number of patient using contraception 12 months post discharge as ascertained by telephone interview.
Pregnancy - 12 months | 12 months
  Number of pregnancies 12 months post discharge as ascertained by telephone interview.

SECONDARY OUTCOMES:
General contraception usage | up to 5 minutes
  Percent of study population using contraception at time of screening
EHR accuracy | up to 5 minutes
  Percentage of patients where the electronic medical record was inaccurate regarding patient's contraception usage
Contraception initiation | up to 1 hour
  Number of patients in the counseling arm who initiated contraception immediately after study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Spielvogel, MD, Principal Investigator — Sutter Health
Locations (1):
- Sutter Medical Center Sacramento, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curtin SC, Abma JC, Ventura SJ, Henshaw SK. Pregnancy rates for U.S. women continue to drop. NCHS Data Brief. 2013 Dec;(136):1-8. PMID 24314113
- [Background] Vahratian A, Barber JS, Lawrence JM, Kim C. Family-planning practices among women with diabetes and overweight and obese women in the 2002 National Survey For Family Growth. Diabetes Care. 2009 Jun;32(6):1026-31. doi: 10.2337/dc08-2105. Epub 2009 Mar 11. PMID 19279299
- [Background] Kaemmerer M, Vigl M, Seifert-Klauss V, Nagdyman N, Bauer U, Schneider KT, Kaemmerer H. Counseling reproductive health issues in women with congenital heart disease. Clin Res Cardiol. 2012 Nov;101(11):901-7. doi: 10.1007/s00392-012-0474-9. Epub 2012 May 15. PMID 22584383
- [Background] Han SN, Van Peer S, Peccatori F, Gziri MM, Amant F; International Network on Cancer, Infertility and Pregnancy. Contraception is as important as fertility preservation in young women with cancer. Lancet. 2015 Feb 7;385(9967):508. doi: 10.1016/S0140-6736(15)60201-X. No abstract available. PMID 25705843
- [Background] Dominick SA, McLean MR, Whitcomb BW, Gorman JR, Mersereau JE, Bouknight JM, Su HI. Contraceptive Practices Among Female Cancer Survivors of Reproductive Age. Obstet Gynecol. 2015 Sep;126(3):498-507. doi: 10.1097/AOG.0000000000000963. PMID 26181090
- [Background] Kendrick J, Sharma S, Holmen J, Palit S, Nuccio E, Chonchol M. Kidney disease and maternal and fetal outcomes in pregnancy. Am J Kidney Dis. 2015 Jul;66(1):55-9. doi: 10.1053/j.ajkd.2014.11.019. Epub 2015 Jan 16. PMID 25600490
- [Background] Hink E, Bolte AC. Pregnancy outcomes in women with heart disease: Experience of a tertiary center in the Netherlands. Pregnancy Hypertens. 2015 Apr;5(2):165-70. doi: 10.1016/j.preghy.2014.12.001. Epub 2015 Jan 5. PMID 25943639
- [Background] Ghaffari N, Srinivas SK, Durnwald CP. The multidisciplinary approach to the care of the obese parturient. Am J Obstet Gynecol. 2015 Sep;213(3):318-25. doi: 10.1016/j.ajog.2015.03.001. Epub 2015 Mar 4. PMID 25747546
- [Background] Chuang CH, Chase GA, Bensyl DM, Weisman CS. Contraceptive use by diabetic and obese women. Womens Health Issues. 2005 Jul-Aug;15(4):167-73. doi: 10.1016/j.whi.2005.04.002. PMID 16051107
- [Background] O'Brien SH, Klima J, Reed S, Chisolm D, Schwarz EB, Kelleher KJ. Hormonal contraception use and pregnancy in adolescents with sickle cell disease: analysis of Michigan Medicaid claims. Contraception. 2011 Feb;83(2):134-7. doi: 10.1016/j.contraception.2010.06.017. PMID 21237338
- [Background] Lee JK, Parisi SM, Schwarz EB. Contraceptive Counseling and Use among Women with Poorer Health. J Womens Health Issues Care. 2013;2(1):103. doi: 10.4172/2325-9795.1000103. PMID 24971372
- [Background] DeNoble AE, Hall KS, Xu X, Zochowski MK, Piehl K, Dalton VK. Receipt of prescription contraception by commercially insured women with chronic medical conditions. Obstet Gynecol. 2014 Jun;123(6):1213-1220. doi: 10.1097/AOG.0000000000000279. PMID 24807345
- [Background] Guth U, Huang DJ, Bitzer J, Moffat R. Unintended pregnancy during the first year after breast cancer diagnosis. Eur J Contracept Reprod Health Care. 2016 Aug;21(4):290-4. doi: 10.1080/13625187.2016.1180678. Epub 2016 May 26. PMID 27227578
- [Derived] Spielvogel R, Stephens RB, Clark R, Guillen M, Hankins A, Parise C. Providing family planning counseling services for women with chronic medical conditions in an inpatient setting: A randomized feasibility trial. Contraception. 2023 Dec;128:110133. doi: 10.1016/j.contraception.2023.110133. Epub 2023 Aug 6. PMID 37549724